CLINICAL TRIAL: NCT03440021
Title: The Effects of Single-dose Administration of a Novel Selective alpha2c Antagonist on Emotional and Cognitive Processing in Healthy Volunteers: an fMRI Investigation
Brief Title: Single-dose Novel Selective alpha2c Antagonist Pharmaco-MRI Study in Healthy Volunteers
Acronym: SNAP_MRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry); University of Oxford (Other)
Responsible Party: Principal Investigator, Prof. Dan J. Stein, Prof., University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 069/2017; N2/19/8/2 (Other: MCC South Africa); DOH-27-0218-5843 (Registry Identifier: SANCTR)
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteer
Keywords: Noradrenalin Agents; Physiological Effects of Drugs; Mood disorders; Behavioral Symptoms
MeSH Terms: conditions — Mood Disorders; Behavioral Symptoms | interventions — ORM-12741

STUDY DESIGN:
Intervention Model Description: High-dosage (60mg), Low-dosage (10mg), Placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dosage (60mg) ORM-12741 (Experimental): 6 x 10 mg ORM-12741 immediate release capsules in a single dose
  Interventions: Drug: ORM-12741
- Low-dosage (10mg) ORM-12741 (Experimental): 1 x 10 mg ORM-12741 immediate release capsules and 5 x placebo capsules in a single dose
  Interventions: Drug: ORM-12741
- Placebo (Placebo Comparator): 6 x placebo capsules in a single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ORM-12741 — Novel selective alpha2c adrenoceptor antagonist
  Arms: High-dosage (60mg) ORM-12741; Low-dosage (10mg) ORM-12741
Drug: Placebo — Identical in appearance to experimental drug, not psycho-active
  Arms: Placebo

SUMMARY:
The aim of the present study is to investigate changes in neural activity (BOLD signal), as measured using fMRI, in brain areas associated with emotional and working memory during task performance after single-dose administration of a novel selective alpha2c adrenoceptor antagonist (ORM-12741) in healthy volunteers. Further, it will be explored whether ORM-12741 affects connectivity between brain areas in rest, as measured using fMRI, and cognitive performance in the sample under investigation.

ELIGIBILITY:
Inclusion Criteria:

* good command of English language
* right handedness
* normal or corrected-to-normal vision

Exclusion Criteria:

* personal history or active presence of psychiatric conditions
* usage of psychotropic medication within the past 3 months
* pregnancy or breast-feeding status
* systolic blood pressure < 90 mmHg or > 140 mmHg at screening visit
* diastolic blood pressure < 50 mmHg or > 90 mmHg at screening visit
* resting heart rate < 45 beats/minute or > 100 beats/minute at screening visit
* active presence of medical condition at physical examination
* history of major traumatic brain injury
* any other contraindication to MRI of the brain
* use of psychoactive substances incl. alcohol in 24 hours prior to test session

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-06 (Actual)

PRIMARY OUTCOMES:
Effect of ORM-12741 on BOLD signal in fMRI of the brain areas associated with emotional memory | 1-1.5 hours post medication intake
Effect of ORM-12741 on BOLD signal in fMRI of the brain areas associated with working memory | 1-1.5 hours post medication intake

SECONDARY OUTCOMES:
Effect of ORM-12741 on connectivity measures between brain areas as measured with BOLD signal in fMRI obtained in a resting state | 1.5-2 hours post medication intake
Effect of ORM-12741 on memory task performance (as measured by accuracy and response latency) | 1-3 hours post medication intake

CONTACTS AND LOCATIONS:
Overall Officials: Dan J. Stein, MD, PhD, Principal Investigator — University of Cape Town
Locations (1):
- UCT Dept. Psychiatry & Mental Health / CUBIC, Cape Town, Western Cape, South Africa